CLINICAL TRIAL: NCT00545181
Title: Recurrent Bacterial Vaginosis (RBV): Efficiency of Metronidazole in Comparison to Metronidazole and Intravaginal Acidifying Gel: A Randomized Investigator-blinded Controlled Trial
Brief Title: Recurrent Bacterial Vaginosis and Vaginal Acidifying Gel Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Responsible Party: David M. Haas, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0612-58 (Study #)
Record Dates: First submitted 2007-10-15; First posted 2007-10-17 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Bacterial Vaginosis
Keywords: bacterial vaginosis; vaginal acidifying gel; recurrence
MeSH Terms: conditions — Vaginosis, Bacterial; Recurrence | interventions — Metronidazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metronidazole plus gel (Experimental): Receive metronidazole plus vaginal gel
  Interventions: Drug: Vaginal acidifying gel (RepHresh)
- Control- metronidazole alone (Active Comparator): Oral Metronidazole antibiotic therapy alone
  Interventions: Drug: Metronidazole control

INTERVENTIONS:
Drug: Vaginal acidifying gel (RepHresh) — placement of vaginal acidifying gel into vagina to restore "normal" vaginal pH.
  Other Names: RepHresh vaginal gel.
  Arms: Metronidazole plus gel
Drug: Metronidazole control — oral metronidazole therapy alone
  Other Names: metronidazole
  Arms: Control- metronidazole alone

SUMMARY:
Bacterial vaginosis (BV) is a common, complex clinical syndrome characterized by alterations in the normal vaginal flora. Bacterial vaginosis has been associated with a variety of adverse health outcomes including endometritis; post-abortion endometritis; nongonococcal, nonchlamydial pelvic inflammatory disease; and an increased risk of acquiring and transmitting HIV infection. In pregnancy, BV is associated with premature rupture of the membranes, chorioamnionitis, amniotic fluid infection, preterm labor, preterm birth, and postpartum endometritis. Several studies have documented increased postpartum complications in the newborn and infants. The etiology of BV is poorly understood but recurrence is quite common despite treatment. Documented recurrence rate of up to 30% within three months are reported. Small studies have shown that adding vaginal acidifying gel to standard antibiotic regimens may reduce recurrence rates of BV. We plan an RCT comparing standard antibiotic therapy to antibiotics plus vaginal acidifying gel. Our hypothesis is that the addition of an acidifying gel will decrease the chance of recurrence of BV within 3 months.

DETAILED DESCRIPTION:
Women with recurrent BV will be randomly assigned to standard care of metronidazole vs metronidazole plus vaginal acidifying gel. Symptoms and presence of BV will be measured at followup.

ELIGIBILITY:
Inclusion Criteria:

1. All women of between 18-50 years of age.
2. Confirmed current diagnosis of BV using Amsel's criteria.
3. Women with at least total 2 confirmed episodes of BV including most recent episode (by Amsel's criteria) within a six month period or at least total three or more in the past twelve months

Exclusion Criteria:

1. Patient who received antibiotic therapy within the past two weeks.
2. Patients who had co-existing gonorrhea or Chlamydia infection
3. Any contraindications or sensitivity to taking the vaginal gel.
4. Allergy to metronidazole
5. Alcoholics or those unable to abstain from alcohol consumption.
6. Pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Haas, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metronidazole + Acidifying Gel (RepHresh): Receive metronidazole plus vaginal acidifying gel
- Metronidazole Alone: Metronidazole antibiotic therapy alone
Period: Overall Study
Arm/Group | Metronidazole + Acidifying Gel (RepHresh) | Metronidazole Alone
Started | 29 | 25
Completed | 29 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metronidazole + Acidifying Gel (RepHresh) | Metronidazole Alone | Total
Number analyzed (Participants) | 29 | 25 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 25 | 54
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.8 (5.8) | 32.4 (6.9) | 31.0 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 25 | 54
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 25 | 54

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Bacterial Vaginosis
Description: Recurrence by either Amsel's or Nugent's criteria. Amsel's criteria are the presence of 3 of 4 of following: 1. homogenous gray-white vaginal discharge, 2. elevated vaginal pH >4.7, 3. presence of at least 20% of vaginal epithelial cells being clue cells on wet prep microscopy, and 4. positive amine odor test on addition of 10% KOH. Nugent's criteria is based on microscopy and bacterial scoring of lactobaccilus, gardnerella, and curved gram-variable rods. A score of at least 7 is indicative of bacterial vaginosis.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Metronidazole + Acidifying Gel (RepHresh) | Metronidazole Alone
Number analyzed (Participants) | 29 | 25
Participants | 7 | 7
Statistical Analysis 1: Comparison: Metronidazole + Acidifying Gel (RepHresh) vs Metronidazole Alone; Test type: Superiority or Other; p = 0.75, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Metronidazole + Acidifying Gel (RepHresh) | Metronidazole Alone
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/25
Other Adverse Events (participants affected / at risk) | 0/29 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No